CLINICAL TRIAL: NCT02951793
Title: Effect of Recent Alcohol, Smoking and Psychotropic Drug Use on Delirium in ICU
Brief Title: Abuse and Addiction in ICU
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jinwoo Lee, Professor, Seoul National University Hospital
Other Study IDs: addiction742
Record Dates: First submitted 2016-10-11; First posted 2016-11-01 (Estimated); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Substance Withdrawal Syndrome
Keywords: intensive care unit; delirium; substance withdrawal
MeSH Terms: conditions — Substance Withdrawal Syndrome; Delirium | interventions — Ethanol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- AUDIT-C > 4: Significant alcohol use within 1 year prior to ICU admission (AUDIT-C>4)
  Interventions: Other: AUDIT-C
- AUDIT-C <=4: No significant alcohol use within 1 year prior to ICU admission (AUDIT-C: equal or less than 4)
  Interventions: Other: AUDIT-C
- Smoking history positive last year: Who smoke cigarette within 1-year prior to ICU admission
  Interventions: Other: Smoking history
- Smoking history negative last year: Who did not smoke cigarette within 1-year prior to ICU admission
  Interventions: Other: Smoking history
- Prior psychotropic medication use - yes: Who used psychotropic medication within 1-year prior to ICU admission
  Interventions: Other: Prior psychotropic medication use
- Prior psychotropic medication use - no: Who did not use psychotropic medication within 1-year prior to ICU admission
  Interventions: Other: Prior psychotropic medication use

INTERVENTIONS:
Other: AUDIT-C — Patients or their proxy/closest family member(s) undergo a comprehensive questionnaire including AUDIT-C about his/her alcohol behavior during last year and will be categorized into two groups: Those with AUDIT-C>4 versus AUDIT-C of 4 or below.
  Other Names: Alcohol Use Disorders Identification Test
  Groups: AUDIT-C <=4; AUDIT-C > 4
Other: Smoking history — Patients or their proxy/closest family member(s) undergo a comprehensive questionnaire including smoking history during last year and will be categorized into two groups: Current smoker versus ex- or never smoker (we also recorded smoking pack-years to distinguish heavy smokers)
  Groups: Smoking history negative last year; Smoking history positive last year
Other: Prior psychotropic medication use — Patients or their proxy/closest family member(s) undergo a comprehensive questionnaire including psychotropic medication use prior admission to ICU and will be categorized into two groups: Those who use psychotropic medication versus those who do not use psychotropic medication.
  Groups: Prior psychotropic medication use - no; Prior psychotropic medication use - yes

SUMMARY:
Investigators are seeking to determine the impact of recent alcohol, smoking or psychotropic drug use prior to intensive care unit (ICU) admission on incidence of delirium and sedation requirements.

Study design: A prospective observational study, in a medical ICU of a tertiary university hospital.

Methods: For all new ICU admissions, a 1-page questionnaire including Alcohol Use Disorders Identification Test (AUDIT-C), smoking history and prior medication use was given to the patient or closest family members.

Delirium was assessed by trained ICU nurses using Intensive Care Delirium Screening Checklist and Richmond Agitation-Sedation Scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are older than 18 years of age
* New patients admitted to medical ICU for the 1st time during their stay in hospital

Exclusion Criteria:

* Had history of stroke or other primary neurologic disease
* GCS ≤ 8 prior to ICU admission
* Transferred from other ICU (except for emergency ICU stay which is limited to less than 36 hours)
* Not registered within 24 hours after admission
* Refused to participate
* If comatous state persists
* Delirium assessment is not possible due to newly developed neurologic disease, such as cerebral infarction
* Medical ICU stay less than 24 hours
* Readmission to medical ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For all new ICU admissions above age of 18 years, except for those who fulfill exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-03; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Delirium during ICU stay | From date of ICU admission until the date of ICU discharge, whichever came first, assessed up to 3 months

SECONDARY OUTCOMES:
ICU length of stay | From date of ICU admission until the date of first documented discharge from ICU or death, whichever came first, assessed up to 3 months
Mortality | From date of ICU admission until the date of death, assessed up to 3 months
  Death in MICU
Maximal doses of dexmedetomidine | From date of ICU admission until the date of first documented discharge from ICU or death, whichever came first, assessed up to 3 months
Cumulative dose of dexmedetomidine | From date of ICU admission until the date of first documented discharge from ICU or death, whichever came first, assessed up to 3 months
  Cumulative dose of dexmedetomidine during the patient's MICU stay
Cumulative dose of midazolam | From date of ICU admission until the date of first documented discharge from ICU or death, whichever came first, assessed up to 3 months
  Cumulative dose of midazolam during the patient's MICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Jinwoo Lee, Professor, Study Chair — Seoul National University Hospital; Jungsil Lee, M.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No